CLINICAL TRIAL: NCT04386005
Title: Continuous Glucose Monitoring in At-Risk Newborns: A Feasibility Study
Brief Title: Continuous Glucose Monitoring in At-Risk Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: DexCom, Inc. (Industry); Children's Miracle Network (Other)
Responsible Party: Principal Investigator, Natalie Allen, Assistant Professor, Pediatrics, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00014068
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Hypoglycemia
Keywords: blood glucose; continuous glucose monitor
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: All participants will have the continuous glucose monitoring device placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Continuous Glucose Monitoring (Experimental): All participants will have the continuous glucose monitoring device placed.
  Interventions: Device: Continuous Glucose Monitoring Device

INTERVENTIONS:
Device: Continuous Glucose Monitoring Device — The Dexcom G7 Glucose Monitoring System (San Diego, CA) reports continuous interstitial blood glucose concentrations every 5 minutes, does not require calibration, and involves only 1 needle stick to place the sensor. The manufacturer recommends that a single sensor may be used for up to 10 days. The Dexcom G7 system is the only FDA approved CGM system for children (age >2 years).
  Other Names: Dexcom G7

SUMMARY:
Hypoglycemia (low blood glucose) is a very common problem in newborns, and has been associated with poor neurodevelopment, cognition, and school performance. At-risk newborns (infants of diabetic mothers [IDM], large [LGA] and small [SGA] for gestational age infants, and late preterm [LPT] infants) undergo a hypoglycemia screening protocol that involves numerous intermittent needle sticks to test glucose levels on bedside glucometers; however, continuous glucose monitoring (CGM, currently not approved for clinical use in babies), via a small sensor placed in the thigh (only 1 needle stick), would likely decrease pain while providing continuous glucose levels. This study will evaluate the feasibility, safety, and precision of CGM in at-risk newborns, and determine if this method would decrease the amount of painful procedures and episodes of hypoglycemia missed by intermittent sampling.

As part of regular medical care, participants will undergo intermittent blood glucose screening with heel sticks as per the current hospital standard of care protocol. Regular medical care involves checking the participant's blood glucose via heel stick every few hours using a bedside glucometer, with another heel stick to confirm low values in the laboratory. If the participant has low values, he/she may be treated with oral glucose gel, feedings of breast milk or formula, or intravenous (IV) fluids in the Neonatal Intensive Care Unit (NICU). This research study involves placing a CGM device in addition to undergoing the current blood glucose screening protocol and treatment.

As soon as possible after birth, a continuous glucose monitoring device (Dexcom G7) will be placed on the participant's thigh by a research team member, and will blindly continuously record glucose levels that will be analyzed after discharge. Everyone who agrees to participate in this study will have placement of this experimental device.

The investigational device will stay in place for the same amount of time that a participant is undergoing blood glucose monitoring as per the current standard of care protocol, for a maximum of 7 days. A participant may need to have his/her blood glucose checked after 7 days for regular medical care (and not for research), because his/her glucose concentrations are still low. Being in the research study will not affect a participant's medical care, and will not affect how long he/she needs blood glucose monitoring or treatment.

A research team member will place and remove the CGM. Nurses will evaluate the site of the device for signs of irritation, infection, bleeding, and any other issues at least 3 times per day. After discharge from the hospital, data will be collected from the participant's medical record and participant's mother's medical record, including the participant's sex and birth weight, blood glucose values, details of feedings, treatments given for low glucose concentrations, and NICU admission data. Data that will be collected from the participant's mother's medical record includes age and race, prenatal data, medical history, and medication use. The participant's parents will be asked to fill out a short survey about their experience with this device when it is removed.

ELIGIBILITY:
Inclusion Criteria:

* At-risk newborns (<48 hours old, all sexes) admitted to the Newborn Nursery or the NICU who meet any of the below criteria:

  1. Infant of a diabetic mother (IDM, pre-existing or gestational diabetes)
  2. Large for gestational age (LGA, >90th percentile [sex-specific])
  3. Small for gestational age (SGA, <10th percentile [sex-specific])
  4. Late preterm (LPT, 34 0/7 to 36 6/7 weeks' gestation)
* Any newborn undergoing routine blood glucose screening in the newborn nursery per the Neonatal Hypoglycemia protocol (includes newborns of mothers taking oral hypoglycemic agents, beta-blocker medications, or systemic steroids within 7 days before delivery; and newborns with clinical manifestations of hypoglycemia)

Exclusion Criteria:

* Birth weight <2kg
* hypoxic-ischemic encephalopathy
* a contraindication to oral feeding
* abnormal skin that will preclude placement of the CGM (e.g., skin on the thigh that is not intact)
* chromosomal abnormalities or severe congenital anomalies identified ante- or postnatally
* infants who are not expected to survive or who are in extremis
* additional risk of immunocompromise, including:

  1. Skin infections, such as staphylococcus or streptococcus skin infections and herpes (skin, eye, and mouth disease) infection
  2. Skin diseases that add additional risk, such as epidermolysis bullosa, ichthyosis, peeling skin syndrome, and hemangiomas
  3. Systemic sepsis, viral syndromes
  4. Immune diseases such as severe combined immunodeficiency, cancer, T-cell or B-cell deficiencies, inborn errors of metabolism, chromosomal abnormalities, glycogen storage diseases, genetic diseases
  5. Abdominal wall defects

Ages: 1 Minute to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Agreement of blood glucose concentrations from CGM vs intermittent monitoring | 1-7 days
  Bland-Altman analysis to evaluate bias and the agreement interval between CGM and intermittent testing
Likert-scale questionnaire results from parents, nurses, and research team | 7 days
  Feasibility of the CGM device will be evaluated by administering Likert-scale questionnaire results from parents, nurses, and research team. Questionnaires will assess acceptability of using the device by parents, nurses, and researchers; and ease of use, placement, and maintenance of the device.
Difference in number of needle sticks with CGM vs intermittent glucose monitoring | 1-7 days
  The total number of estimated needle sticks with GCM will be compared to the total number of needle sticks from intermittent monitoring, using t-test.
Difference in number of episodes of hypoglycemia diagnosed with CGM vs intermittent glucose monitoring | 1-7 days
  Total number of hypoglycemic episodes (blood glucose concentration <40 mg/dL at <4 hours, and <45 mg/dL thereafter) from GCM (episodes lasting >10 minutes) will be compared to the total number of hypoglycemic episodes from intermittent monitoring using t-test. Area under curve analysis will be completed to evaluate duration and severity of hypoglycemic episodes from CGM vs intermittent monitoring, as well as the response to treatment (feedings, dextrose gel, IV dextrose boluses, and dextrose infusions) and timing to normalization of glucose concentrations.

SECONDARY OUTCOMES:
Number of participants with adverse outcomes at the device site | 3 times per day for 1-7 days
  Safety of CGM device will be evaluated by examinations for the presence of irritation, infection, cellulitis, bleeding, or other concerns at the device site.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R. Kaiser, MD, MA, Principal Investigator — Penn State Health Milton S Hershey Medical Center
Locations (1):
- Penn State Health Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Nothing will be shared

REFERENCES:
- [Background] Hay WW Jr, Raju TN, Higgins RD, Kalhan SC, Devaskar SU. Knowledge gaps and research needs for understanding and treating neonatal hypoglycemia: workshop report from Eunice Kennedy Shriver National Institute of Child Health and Human Development. J Pediatr. 2009 Nov;155(5):612-7. doi: 10.1016/j.jpeds.2009.06.044. No abstract available. PMID 19840614
- [Background] Kaiser JR, Bai S, Gibson N, Holland G, Lin TM, Swearingen CJ, Mehl JK, ElHassan NO. Association Between Transient Newborn Hypoglycemia and Fourth-Grade Achievement Test Proficiency: A Population-Based Study. JAMA Pediatr. 2015 Oct;169(10):913-21. doi: 10.1001/jamapediatrics.2015.1631. PMID 26301959
- [Background] Harris DL, Weston PJ, Harding JE. Incidence of neonatal hypoglycemia in babies identified as at risk. J Pediatr. 2012 Nov;161(5):787-91. doi: 10.1016/j.jpeds.2012.05.022. Epub 2012 Jun 23. PMID 22727868
- [Background] Committee on Fetus and Newborn; Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. Pediatrics. 2011 Mar;127(3):575-9. doi: 10.1542/peds.2010-3851. Epub 2011 Feb 28. PMID 21357346
- [Background] Galderisi A, Facchinetti A, Steil GM, Ortiz-Rubio P, Cavallin F, Tamborlane WV, Baraldi E, Cobelli C, Trevisanuto D. Continuous Glucose Monitoring in Very Preterm Infants: A Randomized Controlled Trial. Pediatrics. 2017 Oct;140(4):e20171162. doi: 10.1542/peds.2017-1162. Epub 2017 Sep 15. PMID 28916591
- [Background] Agus MSD, Wypij D, Nadkarni, VM. Tight Glycemic Control in Critically Ill Children. N Engl J Med. 2017 Jun 8;376(23):e48. doi: 10.1056/NEJMc1703642. No abstract available. PMID 28591530
- [Background] Beardsall K, Vanhaesebrouck S, Ogilvy-Stuart AL, Vanhole C, Palmer CR, van Weissenbruch M, Midgley P, Thompson M, Thio M, Cornette L, Ossuetta I, Iglesias I, Theyskens C, de Jong M, Ahluwalia JS, de Zegher F, Dunger DB. Early insulin therapy in very-low-birth-weight infants. N Engl J Med. 2008 Oct 30;359(18):1873-84. doi: 10.1056/NEJMoa0803725. PMID 18971490
- [Background] Shah R, McKinlay CJD, Harding JE. Neonatal hypoglycemia: continuous glucose monitoring. Curr Opin Pediatr. 2018 Apr;30(2):204-208. doi: 10.1097/MOP.0000000000000592. PMID 29346140
- [Background] Stechova K, Cerny M, Brabec R, Ulmannova T, Bartaskova D, Spalova I, Zoban P. Experience with real time continuous glucose monitoring in stabilising fluctuating glycaemia during intensive care of the preterm infant of a diabetic mother. J Matern Fetal Neonatal Med. 2014 Sep;27(13):1389-91. doi: 10.3109/14767058.2013.858686. Epub 2013 Nov 13. PMID 24156750
- [Background] Uettwiller F, Chemin A, Bonnemaison E, Favrais G, Saliba E, Labarthe F. Real-time continuous glucose monitoring reduces the duration of hypoglycemia episodes: a randomized trial in very low birth weight neonates. PLoS One. 2015 Jan 15;10(1):e0116255. doi: 10.1371/journal.pone.0116255. eCollection 2015. PMID 25590334
- [Background] Wackernagel D, Dube M, Blennow M, Tindberg Y. Continuous subcutaneous glucose monitoring is accurate in term and near-term infants at risk of hypoglycaemia. Acta Paediatr. 2016 Aug;105(8):917-23. doi: 10.1111/apa.13479. Epub 2016 Jun 8. PMID 27203555
- [Background] Harris DL, Battin MR, Weston PJ, Harding JE. Continuous glucose monitoring in newborn babies at risk of hypoglycemia. J Pediatr. 2010 Aug;157(2):198-202.e1. doi: 10.1016/j.jpeds.2010.02.003. Epub 2010 Mar 24. PMID 20338573
- [Background] Anand KJ, Coskun V, Thrivikraman KV, Nemeroff CB, Plotsky PM. Long-term behavioral effects of repetitive pain in neonatal rat pups. Physiol Behav. 1999 Jun;66(4):627-37. doi: 10.1016/s0031-9384(98)00338-2. PMID 10386907
- [Background] Patel NS, Duke RP, Tian Z, Zhou S, Kaiser JR. Agreement between intermittent glucose concentrations and continuous glucose monitoring in at-risk newborns. J Perinatol. 2024 Sep;44(9):1367-1368. doi: 10.1038/s41372-024-01906-6. Epub 2024 Feb 19. No abstract available. PMID 38374217
- See also: 5. "Births and Natality." National Center for Health Statistics, Centers for Disease Control and Prevention — http://www.cdc.gov/nchs/fastats/births.htm